CLINICAL TRIAL: NCT00700284
Title: Phase I Study of a Vaginal Ring for Delivery of TMC120 (Dapivirine) as a Vaginal Microbicide
Brief Title: Feasibility Study of a Vaginal Ring for Delivery of TMC120 (Dapivirine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Zeda Rosenberg ScD, International Partnership for Microbicides
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 001, TMC120-C130
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: HIV-I; Reverse transcriptase inhibitors; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: placebo vaginal ring
- B (Experimental)
  Interventions: Drug: TMC120 (dapivirine) vaginal ring

INTERVENTIONS:
Drug: placebo vaginal ring — vaginal ring containing no TMC120 (dapivirine)
  Arms: A
Drug: TMC120 (dapivirine) vaginal ring — vaginal ring containing 120 mg TMC120 (dapivirine)
  Arms: B

SUMMARY:
The purpose of this trial was to evaluate the safety and feasibility of using a vaginal ring to deliver the candidate microbicide TMC120 (dapivirine). Twelve women initially underwent 7-day exposure to a placebo ring containing no investigational agent. They then underwent 7-day exposure to a ring containing 120 mg of TMC120 (dapivirine). Feasibility was assessed in terms of safety and tolerability as well as drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-50 years, inclusive
* Willing and able to provide written informed consent
* HIV-uninfected and otherwise healthy
* Willing to abstain from sexual activity and use of vaginal products while participating in the trial
* Currently using oral contraceptives for pregnancy prevention
* Willing to use oral contraceptives as needed to avoid menstruation while taking part in this trial

Exclusion Criteria:

* History of alcoholism, drug abuse, psychosis, antagonistic personality, poor motivation, or other emotional or intellectual problems that are likely to invalidate the informed consent process or adversely impact compliance with protocol requirements.
* History of allergy to TMC120 or to the constituents of the vaginal ring.
* History of hypersensitivity to propofol, or other contraindication to general anesthesia or sedation
* History of diagnosis of and/or treatment for a sexually transmitted disease within the last three months.
* History of genital tract surgery within the last month
* Currently pregnant or breastfeeding, or within two months of last pregnancy outcome
* Currently or within one month of participating in any other clinical research trial
* Current (during screening) diagnosis of any genital infection
* Current vulvar of vaginal symptoms
* Current non-iatrogenic pelvic/colposcopic exam findings involving deep epithelial disruption

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-10; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of a vaginal ring containing TMC120 (dapivirine) | 7 days
TMC120 (dapivirine) concentrations in vaginal fluids, vaginal and cervical epithelial tissue, and plasma | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Luc Van Bortel, Principal Investigator — Drug Research Unit, UZ Gent
Locations (1):
- Drug Research Unit, UZ Gent, Ghent, Belgium